CLINICAL TRIAL: NCT07246707
Title: A Phase I Clinical Study on the Safety, Tolerability, and Efficacy of KSV01 Injection in Patients With Relapsed/Refractory B-Cell Acute Lymphoblastic Leukemia
Brief Title: KSV01 Injection as the Therapy for Relapsed/Refractory B-Cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: TCRx Therapeutics Co.Ltd (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSV01-R102
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: B-ALL

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KSV01 Injection (Experimental): KSV01 Injection is one kind of third-generation non-replicative self-inactivating lentivirus vector.
  Interventions: Drug: KSV01 Injection

INTERVENTIONS:
Drug: KSV01 Injection — KSV01 Injection is one kind of third-generation non-replicative self-inactivating lentivirus vector.

SUMMARY:
This is a single center, single arm, open-label, dose escalation, phase 1 study to evaluate the safety, tolerability and preliminary efficacy of KSV01 injection for patients with relapsed/refractory B-Cell acute lymphoblastic leukemia (r/r B-ALL).

DETAILED DESCRIPTION:
This investigator-initiated clinical study aims to evaluate KSV01 injection, the third-generation self-inactivating lentiviral vector that carries CD19 CAR, in patients with r/r B-ALL. The study employs a BOIN design to assess safety, tolerability, and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and provision of written informed consent by the patient or their legally authorized representative.
2. Aged 18 to 80 years (inclusive), any gender.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
4. Life expectancy > 3 months.
5. Diagnosis of B-cell Acute Lymphoblastic Leukemia (B-ALL) according to the 2016 WHO classification, with relapsed/refractory disease defined by meeting at least one of the following criteria:

   * Relapse within 12 months of achieving first remission with standard therapy.
   * Primary refractory disease: failure to achieve Complete Remission (CR) after two or more cycles of standard chemotherapy.
   * Relapsed disease after two or more instances of CR.
   * Relapsed or refractory disease following autologous or allogeneic Hematopoietic Stem Cell Transplantation (HSCT).
6. Documented CD19-positive leukemia cells in bone marrow or peripheral blood within 1 month prior to screening.
7. Morphological disease in the bone marrow (blasts ≥5%).
8. For patients with Philadelphia chromosome-positive ALL (Ph+ ALL): must be refractory or intolerant to at least two Tyrosine Kinase Inhibitors (TKIs), including at least one second-generation TKI. Patients with a T315I mutation are exempt from prior TKI salvage therapy.
9. Absolute Lymphocyte Count (ALC) ≥ 100/μL.
10. Adequate organ function as defined by:

    1. Hepatic: Alanine aminotransferase (ALT) ≤ 3 × Upper Limit of Normal (ULN); Aspartate aminotransferase (AST) ≤ 3 × ULN; Total bilirubin ≤ 2 × ULN (or ≤ 3 × ULN with a diagnosis of Gilbert's syndrome, with direct bilirubin ≤ 1.5 × ULN).
    2. Renal: Creatinine clearance (calculated by Cockcroft-Gault formula) ≥ 60 mL/min.
    3. Pulmonary: Oxygen saturation (SaO2) ≥ 92% on room air, and no active pulmonary infection.
    4. Cardiac: Left Ventricular Ejection Fraction (LVEF) ≥ 40% by echocardiography; absence of significant pericardial effusion; no clinically significant electrocardiogram (ECG) abnormalities.
11. For women of childbearing potential: negative urine or serum pregnancy test at screening, and agreement to use effective contraception for at least 1 year post-infusion. Male subjects with partners of childbearing potential must agree to use effective barrier contraception for at least 1 year post-infusion.
12. For subjects with prior blinatumomab (CD3-CD19 bispecific T-cell engager) therapy: CD19 tumor expression on blasts (from bone marrow or peripheral blood) must be documented after the most recent cycle of blinatumomab. If CD19 expression is quantified, the percentage of CD19-positive blasts must be ≥90%.

Exclusion Criteria:

1. Diagnosis of Burkitt's leukemia/lymphoma according to WHO 2016, or chronic myeloid leukemia in accelerated or blast phase.
2. History of another primary malignancy that has not been in continuous remission for at least 2 years. Exceptions to the 2-year limit include: non-melanoma skin cancer, curatively treated Stage I solid tumor with low risk of recurrence, cured carcinoma in situ of the cervix (biopsy-confirmed) or squamous intraepithelial lesion on Pap smear, and cured localized prostate cancer.
3. Uncontrolled active infection within 4 weeks prior to enrollment.
4. Active hepatitis B or hepatitis C virus infection.
5. HIV infection.
6. Positive for Treponema pallidum(syphilis).
7. Severe active autoimmune disease or immunodeficiency, with the exception of well-controlled Type I diabetes and thyroid disorders.
8. History of severe allergy or hypersensitivity to macromolecular biological agents (e.g., antibodies, cytokines).
9. Participation in another interventional clinical trial within 4 weeks prior to enrollment.
10. History of clinically significant central nervous system (CNS) disorders, including but not limited to epilepsy, paresis, aphasia, stroke, severe head injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome.
11. Central Nervous System (CNS) involvement:

    * Presence of CNS 3 disease, defined as detectable blasts in the cerebrospinal fluid (CSF) with ≥5 WBCs/mm³, with or without neurological symptoms.
    * Presence of CNS 2 disease, defined as detectable blasts in the CSF with <5 WBCs/mm³ AND the presence of neurological symptoms.

    Note: Subjects with CNS 1 status (no detectable leukemic blasts in CSF) and subjects with CNS 2 status without significant clinical neurological abnormalities are eligible.
    * History or presence of any CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, any autoimmune disorder involving the CNS, posterior reversible encephalopathy syndrome, or cerebral edema.
12. History of concomitant genetic syndromes associated with bone marrow failure, such as Fanconi anemia, Kostmann syndrome (severe congenital neutropenia), Shwachman-Diamond syndrome.
13. History of any of the following cardiovascular conditions within the past 6 months: New York Heart Association (NYHA) Class III or IV heart failure, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease.
14. Active psychiatric illness.
15. History of drug abuse/addiction.
16. Use of the following medications or therapies:

    1. Salvage systemic therapy (including chemotherapy, TKIs for Ph+ ALL, and blinatumomab) within 1 week or 5 half-lives (whichever is shorter) prior to study drug infusion.

       Note:

       TKIs and hydroxyurea must be discontinued at least 72 hours prior to study drug infusion.* 6-mercaptopurine, 6-thioguanine, methotrexate (standard dose), cytarabine (standard dose), vincristine, and asparaginase must be discontinued at least 1 week prior.* Intrathecal chemotherapy for CNS prophylaxis must be discontinued at least 1 week prior.* PEG-asparaginase must be discontinued at least 4 weeks prior.*
    2. Prior anti-CD19 therapy other than blinatumomab.
    3. History of Grade 4 neurological toxicity (per CTCAE v5.0) or Grade 4 CRS (per Lee 2014 criteria) during prior blinatumomab treatment.
    4. Prior treatment with alemtuzumab within 6 months, or with clofarabine or cladribine within 3 months prior to study drug infusion.
    5. Systemic treatment for Graft-versus-Host Disease (e.g., calcineurin inhibitors, methotrexate, mycophenolate mofetil, sirolimus, thalidomide) or immunosuppressive antibody therapy (e.g., anti-CD20, anti-TNF, anti-IL-6, or anti-IL-6R antibodies) within 4 weeks prior to enrollment.
    6. Any prior systemic therapy with inhibitory/stimulatory immune checkpoint molecules (e.g., ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists). A washout period of at least 3 half-lives from the last dose is required before enrollment.
    7. Radiotherapy: Non-CNS directed radiotherapy within 2 weeks or CNS-directed radiotherapy within 8 weeks prior to study drug infusion.
    8. Corticosteroids: Therapeutic doses of corticosteroids (defined as prednisone equivalent >20 mg/day) within 72 hours prior to study drug infusion. Physiologic replacement doses, and topical or inhaled steroids are permitted.
    9. Prior gene therapy.
    10. Prior adoptive cell therapy.
17. Acute Graft-versus-Host Disease (GVHD) of Grade II to IV per Glucksberg criteria, or overall grade B-D per the IBMTR Severity Index; OR acute or chronic GVHD requiring systemic therapy within 4 weeks prior to enrollment.
18. Administration of a live vaccine within 4 weeks prior to enrollment.
19. Pregnancy or lactation.
20. Any condition that, in the investigator's judgment, may compromise the subject's ability to complete all required study visits and procedures (including follow-up), or comply with the study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity | 28 days after administration
  DLT evaluation period: The DLT evaluation period is defined as within 28 days (inclusive) after the subjects' first administration of KSV01 injection during the dose escalation stage. All adverse events should be graded and evaluated in accordance with CTCAE v5.0. Among them, cytokine release syndrome (CRS) and immune effector cell-related neurotoxicity syndrome (ICANS) should be determined and graded in accordance with the standards of the American Society for Transplantation and Cell Therapy (ASTCT).

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No